CLINICAL TRIAL: NCT07129538
Title: Outcomes of Inspiratory Muscle Training in FMF Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of physical therapy for Cardiovascular, Respiratory disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00014233-32
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Familial Mediterranean Fever
MeSH Terms: conditions — Familial Mediterranean Fever

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMR group (Experimental): Familial mediterranean fever (FMF adolescents ) in this inspiratory muscle retraining group (IMR group) will contain 20 FMF adolescents. IMR group will receive two IMR sessions daily, five times weekly, for eight weeks (every IMR session will contain 3 sets of IMR and the set will contain 10 breath cycles).. also this group will receive their prescribed colchicine medications daily
  Interventions: Other: inspiratory muscle retraining
- control group (Other): Familial mediterranean fever (FMF adolescents ) will be group of FMF will contain 20 FMF adolescents. this group will receive their prescribed colchicine medications daily
  Interventions: Other: colchicine only

INTERVENTIONS:
Other: inspiratory muscle retraining — Familial mediterranean fever (FMF adolescents ) will be inspiratory muscle retraining group (IMR group) that will contain 20 FMF adolescents. IMR group will receive two IMR sessions daily, five times weekly, for eight weeks (every IMR session will contain 3 sets of IMR and the set will contain 10 breath cycles).. this group will receive their prescribed colchicine medications daily
  Arms: IMR group
Other: colchicine only — Familial mediterranean fever (FMF adolescents ) will be collected in this group OF FMF that will contain 20 FMF adolescents. this group will receive their prescribed colchicine medications daily for eight weeks
  Arms: control group

SUMMARY:
Familial mediterranean fever (FMF) is common to be diagnosed before age of 18 . this disorder is connected with deterioration in exercise tolerance, pulmonary capacities, fatigue tolerance,

DETAILED DESCRIPTION:
Familial mediterranean fever (FMF adolescents ) will be collected to be cateogarized to inspiratory muscle retraining group (IMR group) or control waitlist grouping. every group OF FMF will contain 20 FMF adolescents. IMR group will receive two IMR sessions daily, five times weekly, for eight weeks (every IMR session will contain 3 sets of IMR and the set will contain 10 breath cycles).. both groups will receive their prescribed colchicine medications daily

ELIGIBILITY:
Inclusion Criteria:

* FMF adolecents
* ages 13 -17 years
* forty patients

Exclusion Criteria:

* cardiac problems
* renal problems
* liver problems
* diabetes
* brain problems

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — self-representation of gender identity.
Enrollment: 40 (Estimated)
Dates: Start 2025-05-10 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Multidimensional Scale of Fatigue extracted from total score of pediatric quality of life | it will be measured after 8 weeks
  it will assess fatigue perception

SECONDARY OUTCOMES:
cognitive fatigue subscale of Multidimensional Scale of Fatigue related pediatric quality of life | it will be measured after 8 weeks
  it will assess cognitive fatigue perception
sleep and rest fatigue subscale of Multidimensional Scale of Fatigue related pediatric quality of life | it will be measured after 8 weeks
  it will assess fatigue perception during sleep and rest
general fatigue subscale of Multidimensional Scale of Fatigue related pediatric quality of life | it will be measured after 8 weeks
  it will assess general fatigue perception
six minute walk distance | it will be measured after 8 weeks
  it will assess distance covered by FMF patients in six minutes of ongoing walking
Forced vital capacity | it will be measured after 8 weeks
  it is a pulmonary capacity test
Forced exhalation volume (at first second of exhalation) | it will be measured after 8 weeks
  it is a pulmonary function testing
Ration of Forced exhalation volume (at first second of exhalation) to forced exhalation capacity | it will be measured after 8 weeks
  it is a pulmonary function testing
maximum inhalation pressure | it will be measured after 8 weeks
  it is indicator for inspiratory muscular strength
physical sum of child health qestionnaire | it will be measured after 8 weeks
  it is an indiactor for physical quality of life
mental sum of child health qestionnaire | it will be measured after 8 weeks
  it is an indiactor for mental quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Ali MA Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Faculty of physical therapy, Giza, Dokki, Egypt